CLINICAL TRIAL: NCT04348058
Title: Telephone Services for Participation Improvement in Colorectal Cancer Screening: a Randomized Health Services Study
Brief Title: Telephone Services for Participation in Colorectal Cancer Screening
Acronym: ColoPhone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Ministry of Health, Poland (Other Government); Screening up, Poland (Unknown)
Responsible Party: Principal Investigator, Marek Bugajski, PhD, MD, Principal Investigator, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ColoPhone
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Participation Rate, Patient
Keywords: colorectal cancer screening; screening colonoscopy; screening participation; telephone services
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Invitation letter and reminder letter to screening colonoscopy
- Call Center (Experimental): Telephone recruitment by motivational conversation and colonoscopy appointment
  Interventions: Behavioral: Telephone recruitment to screening colonoscopy
- Combined (Experimental): Non responders to invitation and reminder letter will be recruited by telephone conversation
  Interventions: Behavioral: Combined methods recruitment to screening colonoscopy

INTERVENTIONS:
Behavioral: Telephone recruitment to screening colonoscopy — Utilisation of dedicated call center for recruitment to screening program instead of traditional, paper invitation
  Arms: Call Center
Behavioral: Combined methods recruitment to screening colonoscopy — Utilisation of dedicated call center for recruitment to screening program in participants, who did not respond to traditional, paper invitation
  Arms: Combined

SUMMARY:
A multicentre randomized health services study within the population-based primary colonoscopy screening program (PCSP) in Poland. Individuals, aged 55-60 years, willl be randomized in a 1:1:1 ratio to arms: (1) Invitation by post, (2) Call Center or (2) Combined invitation methods. The primary outcome measure is rate of participation in screening colonoscopy. The sample size of 6 300 participants will detect 3 to 5 percentage point differences (depending on the arms comparison) in participation rate between groups with 80% power and significance level 0.05, using Ochran-Mantel-Haenszel test.

DETAILED DESCRIPTION:
This randomized health services study will be performed within national population-based screening program (PCSP) in Poland, including its population, infrastructure and database system.

Individuals aged 55-64 years old, included in PCSP willl be randomly assigned (in 1:1:1 ratio, stratified by gender, age, place of residence) to study arms and invited to screening colonoscopy to local PSCP centers.

Invitation process by post in Control group (1) and partially in Combined group (3) - will be performed by coordinating PCSP center (practice as usual).

Recruitment by telephone conversation in Call Center group (2) and partially in Combined group (3) - will be performed by Screening Up call center company. Colonoscopies will be performed in 6 selected PCSP centers.

The sample size of 2,100 participants per group (350 participants from each group in each center, assuming 5% drop out and access to telephone numbers of 30% participants in relevant arms; calculation is based on a 95% confidence interval +/- 5% error probability) was calculated to detect a difference in participation rate of 15% in control group (based on PCSP participation rate in 2019) vs. 18.7% in Call Center group vs 25% in Combined Invitation group (0.025 significance level with 80% power). The difference was calculated for the Cochran-Mantel-Haenszel test, assuming that the initial reporting in the control group will be as high as it was in 2019.

Differences in participation rate to screening colonoscopy between the study groups and the control group will be performed using Ochran-Mantel-Haenszel test (two-sided analysis), taking into account initial differences between rates at the significance level of 0.05.

The Principal Investigator of the study asked the Bioethical Committee with a request to release participants from signing of informed consent form to participation in the study, as they take part in a nationwide PSCP, financed by Ministry of Health in Poland - the study character is the Randomized Health Services Study.

ELIGIBILITY:
Inclusion Criteria:

* population included to invitation within Polish population based Colorectal cancer Screening Program (PCSP)

  * 55-64 of age
  * no history of CRC
  * no history of screening colonoscopy within PCSP
* adress of residence near (not further than 40 kilometers) local PCSP centers (selected for the study based on population density)

Exclusion Criteria:

* none

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6300 (Estimated)
Dates: Start 2020-08-20 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Participation rate to screening colonoscopy within PCSP per recruitment strategy | 26 weeks after intervention
  The percentage of study participants who underwent screening colonoscopy relative to all PCSP participants to whom the invitation was sent in a given group during the observation period (intention-to-screen analysis)

SECONDARY OUTCOMES:
Response rate to invitation to screening colonoscopy | 26 weeks after intervention
  Contact with local PCSP center

CONTACTS AND LOCATIONS:
Locations (1):
- The Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Mazovian, Poland

REFERENCES:
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] European Colorectal Cancer Screening Guidelines Working Group; von Karsa L, Patnick J, Segnan N, Atkin W, Halloran S, Lansdorp-Vogelaar I, Malila N, Minozzi S, Moss S, Quirke P, Steele RJ, Vieth M, Aabakken L, Altenhofen L, Ancelle-Park R, Antoljak N, Anttila A, Armaroli P, Arrossi S, Austoker J, Banzi R, Bellisario C, Blom J, Brenner H, Bretthauer M, Camargo Cancela M, Costamagna G, Cuzick J, Dai M, Daniel J, Dekker E, Delicata N, Ducarroz S, Erfkamp H, Espinas JA, Faivre J, Faulds Wood L, Flugelman A, Frkovic-Grazio S, Geller B, Giordano L, Grazzini G, Green J, Hamashima C, Herrmann C, Hewitson P, Hoff G, Holten I, Jover R, Kaminski MF, Kuipers EJ, Kurtinaitis J, Lambert R, Launoy G, Lee W, Leicester R, Leja M, Lieberman D, Lignini T, Lucas E, Lynge E, Madai S, Marinho J, Maucec Zakotnik J, Minoli G, Monk C, Morais A, Muwonge R, Nadel M, Neamtiu L, Peris Tuser M, Pignone M, Pox C, Primic-Zakelj M, Psaila J, Rabeneck L, Ransohoff D, Rasmussen M, Regula J, Ren J, Rennert G, Rey J, Riddell RH, Risio M, Rodrigues V, Saito H, Sauvaget C, Scharpantgen A, Schmiegel W, Senore C, Siddiqi M, Sighoko D, Smith R, Smith S, Suchanek S, Suonio E, Tong W, Tornberg S, Van Cutsem E, Vignatelli L, Villain P, Voti L, Watanabe H, Watson J, Winawer S, Young G, Zaksas V, Zappa M, Valori R. European guidelines for quality assurance in colorectal cancer screening and diagnosis: overview and introduction to the full supplement publication. Endoscopy. 2013;45(1):51-9. doi: 10.1055/s-0032-1325997. Epub 2012 Dec 4. PMID 23212726
- [Background] Rex DK, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Levin TR, Lieberman D, Robertson DJ. Colorectal Cancer Screening: Recommendations for Physicians and Patients From the U.S. Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2017 Jul;153(1):307-323. doi: 10.1053/j.gastro.2017.05.013. Epub 2017 Jun 9. PMID 28600072
- [Background] Kaminski MF, Kraszewska E, Rupinski M, Laskowska M, Wieszczy P, Regula J. Design of the Polish Colonoscopy Screening Program: a randomized health services study. Endoscopy. 2015 Dec;47(12):1144-50. doi: 10.1055/s-0034-1392769. Epub 2015 Oct 30. PMID 26517847
- [Background] Camilloni L, Ferroni E, Cendales BJ, Pezzarossi A, Furnari G, Borgia P, Guasticchi G, Giorgi Rossi P; Methods to increase participation Working Group. Methods to increase participation in organised screening programs: a systematic review. BMC Public Health. 2013 May 13;13:464. doi: 10.1186/1471-2458-13-464. PMID 23663511
- [Background] Goodwin BC, Ireland MJ, March S, Myers L, Crawford-Williams F, Chambers SK, Aitken JF, Dunn J. Strategies for increasing participation in mail-out colorectal cancer screening programs: a systematic review and meta-analysis. Syst Rev. 2019 Nov 4;8(1):257. doi: 10.1186/s13643-019-1170-x. PMID 31685010